CLINICAL TRIAL: NCT04590300
Title: Impact Des Performances Cognitives et métacognitives Sur l'Apprentissage de Connaissances Lors de la réalisation de Programmes d'éducation thérapeutique
Brief Title: Impact of Cognitive & Metacognitive Performance on Knowledge Learning When Conducting Therapeutic Education Programs
Acronym: MetaCOGNITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00980-39
Record Dates: First submitted 2020-09-10; First posted 2020-10-19 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia (Other): 1 questionnaire at the beginning of the study, before FTE program
  1 questionnaire at the end of FTE
  Interventions: Other: QUESTIONNAIRES
- Bipolar disorder (Other): 1 questionnaire at the beginning of the study, before FTE program
  1 questionnaire at the end of FTE
  Interventions: Other: QUESTIONNAIRES

INTERVENTIONS:
Other: QUESTIONNAIRES — 1 questionnaire at the beginning of the study, before FTE program
  1 questionnaire at the end of FTE

SUMMARY:
People with schizophrenia and bipolar disorder display alterations in cognition and metacognition. These alterations may have an impact on learning during therapeutic education programs.

DETAILED DESCRIPTION:
Patient Therapeutic Education (FTE) is defined as a practice to help patients to acquire or maintain the skills needed to best manage their lives with a chronic disease. FTE includes organized awareness, information, learning and psychological and social assistance about the disease, prescribed treatments, various treatments offered, as well as information on organization of the global health system, and health behaviours. Performed by health professionals trained in this practice, FTE is intended to help patients and their close relatives and to understand their pathology, their treatments, collaborate with health care teams, and maintain or improve their quality of life. It aims to produce a complementary therapeutic effect of other health care interventions

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the study,
* Suffering from a chronic condition for which an therapeutic patient education (TEP) program is proposed.
* Mastering the French language.
* Be a beneficiary of health insurance

Exclusion Criteria:

* Poor understanding of instructions that make it impossible to consent or assess
* Neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of cognitive impairments on knowledge acquired through a therapeutic education program with Montreal Cognitive Assessment (MoCA) | 1 year
  assess the impact of possible cognitive impairments on knowledge acquired through a therapeutic education program Minimum value = 0 & Maximum value = 30 Score < 26 is considered as abnormal
Evaluation of metacognitive impairments on knowledge acquired through a therapeutic education program with Subjective Scale To Investigate Cognition in Schizophrenia (SSTICS) | 1 year
  assess the impact of possible metacognitive impairments on knowledge acquired through a therapeutic education program Minimum value 21

SECONDARY OUTCOMES:
assess the impact of self esteem acquired through a therapeutic education program with Rosenberg scale | 1 year
  assess the evolution in self-esteem following this program.
assess the impact of level of anxiety, acquired through a therapeutic education program with State-Trait-Anxiety Inventory (Forme Y) (STAI-Y) questionnaire | 1 year
  assess the evolution in level of anxiety following this program.
assess the impact of depressive symptomatology acquired through a therapeutic education program with Center for Epidemiologic Studies-Depression (CES-D) scale | 1 year
  assess the evolution in depressive symptoms following this program.
assess the impact of literacy on knowledge acquired through a therapeutic education program with Rapid Estimate for Adult Literacy in Medicine (REALM-R) questionnaire | 1 year
  assess the evolution in quality of life following this program.

CONTACTS AND LOCATIONS:
Overall Officials: Clelia QUILES, MD, Principal Investigator — CH Charles Perrens
Locations (1):
- Centre Hospitalier CHARLES PERRENS, Bordeaux, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xia J, Merinder LB, Belgamwar MR. Psychoeducation for schizophrenia. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD002831. doi: 10.1002/14651858.CD002831.pub2. PMID 21678337
- [Background] Soo SA, Zhang ZW, Khong SJ, Low JEW, Thambyrajah VS, Alhabsyi SHBT, Chew QH, Sum MY, Sengupta S, Vieta E, McIntyre RS, Sim K. Randomized Controlled Trials of Psychoeducation Modalities in the Management of Bipolar Disorder: A Systematic Review. J Clin Psychiatry. 2018 May/Jun;79(3):17r11750. doi: 10.4088/JCP.17r11750. PMID 29727072
- [Background] Flavell J.H. Metacognition and cognitive monitoring. A new area of cognitive-developmental inquiry. Am Psychol. 1979; 34(10):906-11